CLINICAL TRIAL: NCT06192914
Title: Prospective Survey of the Repeated Occurrence of Anaphylactic Reactions in Patients with Food Allergies
Brief Title: EPAP, Interviewstudy
Status: Recruiting | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Margitta Worm, Prof. Dr., Charite University, Berlin, Germany
Other Study IDs: EPAP; EA2/137/21 (Other: local ethic committee)
Record Dates: First submitted 2023-12-11; First posted 2024-01-05 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Food Allergy; Food Allergy Peanut; Allergy; Anaphylactic Shock
Keywords: Food Allergy; Repetitive Reactions; Quality of Life
MeSH Terms: conditions — Food Hypersensitivity; Peanut Hypersensitivity; Hypersensitivity; Anaphylaxis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Food Anaphylaxis Patients: Patients with anaphylaxis to legumes, tree nuts, seeds, cereals and pseudocereals within the last 12 months

SUMMARY:
The goal of this observational study is to learn about repetitive anaphylactic reactions in food allergic patients and to compare the frequency of repetitive reactions between different elicitors in food allergic patients. The main question it aims to answer are:

• Is there an elicitor specific difference in the occurrence of anaphylactic reactions once the elicitor has been identified and the patient received counselling about its avoidance?

Participants will answer questionnaires via a link they will receive via e-mail at baseline and 3, 6, 12 and 24 months after inclusion in the study.

DETAILED DESCRIPTION:
The aim of the study is to establish a cohort of patients who were included in the anaphylaxis registry with an anaphylactic reaction to legumes, tree nuts, seeds, grains or pseudocereals within the previous twelve months. Patients are requested to provide information about the occurrence of new allergic reactions at defined time-points over a period of two years (at baseline, 3, 6, 12, and 24 months). In addition, their eating behavior and the food allergy-specific quality of life will be captured. The investigators intend to track self-management in dealing with anaphylaxis, especially the use of emergency medication. It is examined whether patients react again and whether these are reactions to a known or previously unknown allergen to the patient. By recording the symptoms, it will be checked whether there are certain reaction patterns to specific foods or whether these are patient specific. In addition, the influence of the previous anaphylactic reaction and knowledge of the existing allergy on quality of life, dietary behavior and the ability to use emergency medication should be examined.

This is intended to help improve the care for future patients in order to minimize the risk of repeat reactions.

ELIGIBILITY:
Inclusion Criteria:

* anaphylactic reaction to peanuts, other legumes, tree nuts, seeds (e.g. sesame seed, sunflower seed), cereals (e.g. wheat, oat) or pseudocereals (e.g. quinoa)
* participation in the European Anaphylaxis Registry (Clinical Trials Identifier: NCT05210543)
* possibility and consent to receive links to the follow-up electronic surveys via e-mail and fill out the questionnaires electronically

Exclusion Criteria:

* if inclusion criteria are fulfilled there are no further exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of patients (age 18 years or older) or their parents (patients age 0-17 years). Eligible patients have suffered at least one anaphylactic reaction to peanuts, other legumes, tree nuts, seeds (e.g. sesame seed, sunflower seed), cereals (e.g. wheat, oat) or pseudocereals (e.g. quinoa) within 12 months prior to presentation in a specialised food allergy center that is participating in the European Anaphylaxis Registry and in addition the EPAP follow-up project. If the patient or their parents agree to participate in the European Anaphylaxis Registry and fulfill the other inclusion criteria, they can also participate in the follow up study. We aim to include 322 patients.
Sampling Method: Non-Probability Sample
Enrollment: 322 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2029-02-28 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Frequency of allergic reactions in tree nut and peanut allergic patients within the observation period of the study | 2 years
  The aim is to identify whether the frequency of allergic reactions after the identification of the elicitor of the initial allergic reaction differs between peanuts and tree nuts

SECONDARY OUTCOMES:
Frequency of allergic reactions among patients with different food allergens within the observation period of the study | 2 years
  The aim is to identify whether the frequency of allergic reactions after the identification of the elicitor of the initial allergic reaction differs between different food allergens
The association of food allergy related quality of life, measured via the Food Allergy Quality of Life Questionnaire, with repetitive allergic reactions | 2 years
  An anaphylactic reaction to food can impact quality of life. The investigators want to observe the food allergy related quality of life over the study period and examine whether the existence of repetitive reaction influences quality of life. Food allergy related quality of life is measured via the Food Allergy Quality of Life Questionnaire (FAQLQ). Patients can achieve 1 - 7 points, where a higher score represents a higher impairment of quality of life and 1 point represents no impairment.
The association of eating habits (e.g. frequency of eating out) and the occurrence of repetitive allergic reactions | 2 years
  An anaphylactic reaction to food can influence eating habits and specific eating habits can be related to more frequent accidental allergic reactions. The investigators want to observe whether the eating habits differ between patients with and without recurrent allergic reactions.
  The eating habits are captured with a non-validated questionnaire. Patient are requested to answer, whether they follow a specific diet (e.g. vegan, vegetarian, religious diets) and how often they use specific ways of eating out (e.g. in a restaurant or eating at a friends place). The eating habits are captured at every time point of the study (baseline, 3, 6, 12, 24 months).
Use of emergency medication during a repetitive reaction | 2 years
  The prescripton of emergency medications and the instruction about their use enables patients or their relatives to take care of the primary treatment of anaphylactic reactions. The investigators want to compare whether the use of emergency medication during subsequent anaphylactic reactions increases. Patients are requested to provide details about the use of emergency medication for each allergic reaction they report via the study period.
Use of adrenaline as first line treatment | 2 years
  The instruction about adrenaline autoinjectors and their use as first line treatment in case of an allergic reaction increases the frequency of its use. The investigators want to compare whether the use of adrenaline as a first line treatment during subsequent anaphylactic reactions increases. Patients are requested to provide details about the use of adrenaline for each allergic reaction they report via the study period.
The association of dietary counselling and successful allergen avoidance | 2 years
  The investigators hypothesize that dietary counselling enables patients to avoid their allergen effectively and reduces the number of allergic reactions compared to the time before dietary counselling. Patients are requested to provide the number of allergic reactions throughout the two years before inclusion in the study in the baseline questionnaire. This number will be compared with the number of reactions patients report during the study. The study inclusion always takes place in a specialized allergy center, where every patient receives counselling about allergen avoidance.

CONTACTS AND LOCATIONS:
Overall Officials: Margitta Worm, MD, Principal Investigator — Allergy and Immunology, Department of Dermatology, Venerology and Allergy, Charité Universitätsmedizin Berlin
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, State of Berlin, Germany

IPD SHARING:
Plan to Share IPD: No